CLINICAL TRIAL: NCT04104334
Title: Evaluation of the Impact of Combined Intraoperative Monitoring of Depth of Analgesia, Depth of Anesthesia and Continuous Hemodynamic Data on the Patients Recovery After Cytoreduction Surgery and Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Impact of an Optimised Monitored Anesthesia on the Patients' Recovery After Cytoreduction Surgery Plus HIPEC
Acronym: CHIPNOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in surgical practice and chemotherapy treatment by the surgery team
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, MD, PhD, Professor, Director of Research, Department of Anesthesiology and Pain Medicine of Maisonneuve-Rosemont Hospital, CIUSSS de l'Est de l'Ile de Montreal (CEMTL), Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-1788
Record Dates: First submitted 2019-07-16; First posted 2019-09-26 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Hyperthermia; Colorectal Neoplasms; Oxaliplatin
Keywords: Cytoreduction; HIPEC; Oxaliplatin; Colorectal; Peritoneal; Carcinomatosis; Monitoring; Anesthesia
MeSH Terms: conditions — Hyperthermia; Colorectal Neoplasms; Carcinoma | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 2 groups of patients. Randomization into Monitored group "M" (BIS + NOL + Flotrac EV1000) vs control group "C" (standard of care anesthesia) according to randomization list for a total number of 80 patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization into Monitored group "M" (BIS + NOL + Flotrac EV1000) vs control group "C" (standard of care anesthesia) will be done prior to the entrance in the OR, the day of the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitored group "M" (optimized controlled anesthesia) (Active Comparator): Patients in the Monitored group "M", the NOL index will guide the administration of remifentanil to keep the index between 5-25, and the desflurane will be titrated to keep a BIS index between 45 and 55. Cardiac output and stroke volume variation will be measured by the Flotrac EV1000 system. Patients will receive 250ml fluid challenges with a recommended solution as required, in order to achieve a maximal value of stroke volume.
  Interventions: Drug: Remifentanil infusion, desflurane titration and fluid infusion will be guided by NOL index, BIS index and Flotrac EV1000 system respectively
- Control group "C" (standard of care anesthesia) (Active Comparator): Patients in the Control group "C" will be managed by clinical staff according to usual practice, desflurane will be administered to keep MAC at 1, and remifentanil infusion rate will be adapted to the mean arterial blood pressure to keep it between 65 and 100.
  Interventions: Drug: Remifentanil infusion and desflurane titration will be guided by anesthesia usual practices

INTERVENTIONS:
Drug: Remifentanil infusion, desflurane titration and fluid infusion will be guided by NOL index, BIS index and Flotrac EV1000 system respectively — NOL index will guide the administration of remifentanil to keep the index between 5-25, and the desflurane will be titrated to keep a BIS index between 45 and 55. Cardiac output and stroke volume variation will be measured by the Flotrac EV1000 system. Patients will receive 250ml fluid challenges with a recommended solution as required, in order to achieve a maximal value of stroke volume
  Other Names: Monitoring group
  Arms: Monitored group "M" (optimized controlled anesthesia)
Drug: Remifentanil infusion and desflurane titration will be guided by anesthesia usual practices — Desflurane will be administered to keep MAC at 1, and remifentanil infusion rate will be adapted to the mean arterial blood pressure to keep it between 65 and 100, according to anesthesia usual practices
  Other Names: Control group
  Arms: Control group "C" (standard of care anesthesia)

SUMMARY:
The objective of our PILOT study is to evaluate the impact of a controlled (monitored) randomized anesthesia during cytoreductive surgery with HIPEC to oxaliplatin in order to treat adenocarcinomas of colorectal origin. The combination of NOL monitoring, BIS monitoring and continuous hemodynamic monitoring (FloTrac EV1000 system) can improve patient safety by reducing the length of hospital stay by decreasing total hypnotic doses and intraoperative opioids and side effects following anesthesia.

DETAILED DESCRIPTION:
Title: Evaluation of the combined intraoperative monitoring of depth of analgesia (NOL), depth of anesthesia (BIS) and continuous hemodynamic data (Flotrac EV1000 system) on the patients' recovery after cytoreduction surgery and hyperthermic intraperitoneal chemotherapy (HIPEC). A pilot study.

Hypothesis: Investigators hypothesize that the intraoperative combination of new monitors, NOL index for depth of analgesia, BIS index for depth of anesthesia and Flotrac EV1000 system as continuous hemodynamic monitoring, to guide the delivery of opioids, hypnotics, fluids and inotropes, respectively, will improve the quality of recovery as well as the safety after anesthesia in patients undergoing HIPEC (Hyperthermic Intraperitoneal Chemotherapy) surgery.

Background: so far, only vital signs (mostly, blood pressure and heart rate) helped the anesthesiologist to administer hypnotics agents, analgesics, fluids and inotrope. Many devices have offered pain monitoring for anesthetized patients. The NOL index, a nociception monitor using a multiparametric approach, has shown an excellent sensitivity and specificity in detecting noxious stimuli under general anesthesia. More recently, it has been shown a strong inverse correlation between NOL index response to nociceptive stimulus and the increasing doses of opioid analgesia during surgery. Studies on post-operative outcomes when using intraoperative NOL monitoring to adapt nociception/anti-nociception balance during general anesthesia (GA) also reported in our center an improvement of the time to extubation and of the postoperative recovery criteria in PACU after colorectal surgery in the monitored group, leading to a quicker discharge from PACU (presented as an abstract at ASA 2018; manuscript in preparation). Recent studies also showed that avoiding too deep anesthesia by using the BIS index would improve patients' outcome in terms of morbi-mortality. It is also accepted that intra-venous fluid and inotropic/vasopressor drugs have an important effect on intra and postoperative patients' outcomes, in particular following major gastrointestinal surgery. The use of hemodynamic therapy management algorithms has been recommended in a report commissioned by the Centers for Medicare and Medicaid Services in the USA, and by the National Institute for Health and Care Excellence (NICE) in the UK as well as many groups working in ERAS protocols in Canada (and especially Montreal, McGill University) and worldwide.

Based on our recent systematic review (in preparation) and out of the 69 selected published articles, there is no study so far evaluating precisely the impact of anesthesia on postoperative outcomes, and no study combining the NOL, the BIS indexes and the Flotrac EV1000 system to evaluate the impact of a more precise anesthesia management on the postoperative outcomes after cytoreduction and HIPEC for peritoneal carcinomatosis of colorectal origin. Thus, the idea to propose the present study.

Specific Objectives: primary objective: to compare the time to reach the readiness for discharge from hospital and the total postoperative in-hospital length of stay between the Monitored group "M" (optimized, personalized and controlled anesthesia) versus the control group "C" (standard of care anesthesia). Secondary objectives: to evaluate the quality of recovery from anesthesia in the PACU and on the wards and all the adverse events every day and until patient's discharge from hospital. The emergence and extubation time of patients after anesthesia, time spent in PACU (Aldrete score), intra- and postoperative opioid requirements, pain scores (NRS) for several postoperative days, patients' postoperative recovery and satisfaction (the Quality of Recovery: QOR-15, 6min walking test, MOCA, etc.) will be also compared between the 2 groups. Finally, biological outcomes such as blood gas analysis, serum electrolytes, creatinine, DFG, hemoglobin, white blood cell and platelet counts, CRP, serum albumin, INR, PTT will be evaluated on a standard basis in both the groups.

Methods: 80 patients scheduled for HIPEC surgery with oxaliplatin for bowel adenocarcinoma surgery (without digestive resection) will be included. Randomisation will occur after the participant has provided informed consent and shortly before the surgical procedure is due to start. Patients in the Control group "C" will be managed by clinical staff according to usual practice, desflurane will be administered to keep MAC at 1, and remifentanil infusion rate will be adapted to the mean arterial blood pressure to keep it between 65 and 100. In the Monitored group "M", the NOL index will guide the administration of remifentanil to keep the index between 5-25, and the desflurane will be titrated to keep a BIS index between 45 and 55. Cardiac output and stroke volume variation will be measured by the Flotrac EV1000 system. Patients will receive 250ml fluid challenges with a recommended solution as required, in order to achieve a maximal value of stroke volume. Intraoperative epidural analgesia will be the same for all. Postoperative analgesia will be based on PCEA and hydromorphone for all. All anesthesia related side effects and quality of analgesia and rehabilitation will be evaluated daily and until patient's discharge from hospital.

Data Analysis: all data collected will be analyzed using an intent-to-treat approach. Summary statistics for each group, treatment effects, 95% confidence intervals, and p-values will be presented for primary and secondary outcomes, and process measures. Intraoperative data in the "M" and "C" groups will be compared using parametric (e.g. Student t-test) or non-parametric tests (e.g. Mann-Withney U test, Chi-squared test) depending on type of variables and distribution. General linear models will be used to carry out group comparisons on data on length of hospital stay. Potential pitfalls: analyses for secondary objectives may not be sufficiently powered but will nevertheless provide useful information for designing and conducting a future multicentric study. Bonferroni corrections will be used to protect against type I error.

Significance/Importance: Adding the NOL, the BIS and continuous hemodynamic monitoring will very likely reduce the total length of stay, and improve the postoperative speed and quality of recovery as well as will likely reduce the incidence of complications after cytoreduction + HIPEC procedures.

Study Design: Prospective, randomized controlled study.

Subject Population: Adult patients scheduled to undergo laparotomy for cytoreduction surgery + HIPEC for peritoneal carcinomatosis of colorectal origin and under general anesthesia with an active intraoperative epidural analgesia.

Sample Size: 80 patients will be evaluated in this study.

Study Duration: 2 year(s)

Study Center: Maisonneuve-Rosemont Hospital, Departments of Anesthesiology and Pain Medicine and Department of General Oncologic Surgery, CIUSSS de l'Est-de-l'Île-de-Montreal, Montreal, Quebec, Canada

Adverse Events: None expected.

Subvention/support: Department of Anesthesiology and Pain Medicine of HMR/CEMTL.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II or III
* Patients older than 18 years
* HIPEC for bowel surgery with oxaliplatin + dextrose 5% for a duration of 30 min
* Duration and type of surgery requiring an epidural analgesia via an epidural catheter placed and tunnelled prior the general anesthesia induction and an arterial line placed after induction of general anesthesia.

Exclusion Criteria:

* Any allergy to one drug used in our anesthesia or HIPEC protocol
* Any contra-indication or patient's refusal for epidural placement
* Chronic arrhythmic cardiac conditions
* Chronic pain with use of opioids more than 3 times per week for 4 weeks
* Bowel occlusion
* Physical/mental incapacities
* Unexpected difficult airway requesting excessive, possibly painful airway manipulations.
* Epidural failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The hospital length of stay in days | Evaluated 24 hours postoperative and everyday until hospital discharge, up to 21 days
  The length of hospital stay in group "M" versus group "C" will be evaluated with the readiness for discharge from hospital criteria.
  These criteria for hospital discharge will be precisely and daily evaluated based on the previous published literature from experts who reached a consensus (J.F. Fiore et al. Disease of the Colon and Rectum, volume 55: 4, 2012).
  After these criteria are achieved, discharge may take place.
Tolerance of oral intake | Evaluated 24 hours postoperative and everyday until hospital discharge, up to 21 days
  The length of hospital stay in group "M" versus group "C" will be evaluated with the readiness for discharge from hospital criteria.
  These criteria for hospital discharge will be precisely and daily evaluated based on the previous published literature from experts who reached a consensus (J.F. Fiore et al. Disease of the Colon and Rectum, volume 55: 4, 2012) and this will include:
  - Tolerance of oral intake.
  After these criteria are achieved, discharge may take place.
Recovery of lower gastrointestinal function | Evaluated 24 hours postoperative and everyday until hospital discharge, up to 21 days
  The length of hospital stay in group "M" versus group "C" will be evaluated with the readiness for discharge from hospital criteria.
  These criteria for hospital discharge will be precisely and daily evaluated based on the previous published literature from experts who reached a consensus (J.F. Fiore et al. Disease of the Colon and Rectum, volume 55: 4, 2012) and this will include:
  - Recovery of lower gastrointestinal function.
  After these criteria are achieved, discharge may take place.
Adequate pain control with oral analgesia | Evaluated 24 hours postoperative and everyday until hospital discharge, up to 21 days
  The length of hospital stay in group "M" versus group "C" will be evaluated with the readiness for discharge from hospital criteria.
  These criteria for hospital discharge will be precisely and daily evaluated based on the previous published literature from experts who reached a consensus (J.F. Fiore et al. Disease of the Colon and Rectum, volume 55: 4, 2012) and this will include:
  - Adequate pain control with oral analgesia.
  After these criteria are achieved, discharge may take place.
Ability to mobilize and self-care | Evaluated 24 hours postoperative and everyday until hospital discharge, up to 21 days
  The length of hospital stay in group "M" versus group "C" will be evaluated with the readiness for discharge from hospital criteria.
  These criteria for hospital discharge will be precisely and daily evaluated based on the previous published literature from experts who reached a consensus (J.F. Fiore et al. Disease of the Colon and Rectum, volume 55: 4, 2012) and this will include:
  - Ability to mobilize and self-care.
  After these criteria are achieved, discharge may take place.
Clinical examination and laboratory tests show no evidence of complications or untreated medical problems | Evaluated 24 hours postoperative and everyday until hospital discharge, up to 21 days
  The length of hospital stay in group "M" versus group "C" will be evaluated with the readiness for discharge from hospital criteria.
  These criteria for hospital discharge will be precisely and daily evaluated based on the previous published literature from experts who reached a consensus (J.F. Fiore et al. Disease of the Colon and Rectum, volume 55: 4, 2012) and this will include:
  - Clinical examination and laboratory tests show no evidence of complications or untreated medical problems.
  After these criteria are achieved, discharge may take place.

SECONDARY OUTCOMES:
Intraoperative anesthetic gas' consumption in ml/kg/h | Intraoperative
  Total consumption and absorption of desflurane in ml/kg/h during surgery and for each hour of surgery
Intraoperative remifentanil consumption in mcg/kg/min | Intraoperative
  Total consumption of i.v. remifentanil during surgery and for each hour of surgery
Intraoperative fluid's consumption in ml/h | Intraoperative
  Total of fluid perfused during surgery and for each hour of surgery
Intraoperative number of hypotensive events | Intraoperative
  Total number of hypotensive events during surgery (defined as mean blood pressure below 60)
Intraoperative phenylephrine consumption in mcg/kg/min | Intraoperative
  Total doses of intraoperative infused i.v. phenylephrine and doses per hour
Intraoperative epidural consumption in 3 ml/h | Intraoperative
  Total doses of intraoperative Epidural infusion (lidocaine 2%+epinephrine) and doses per hour
Time for awakening in seconds | Intraoperative
  Time for awakening (eyes opening) at the end of the surgery. Elapsed time in seconds between stopping the gas and opening the eyes of the patient
Time for extubation in seconds | Intraoperative
  Time for extubation in seconds. Elapsed time in seconds between stopping the gas and patient's extubation
Time for transfert to the PACU in seconds | Intraoperative
  Time for transfert to the PACU (Post Anesthesia Care Unit) in seconds, after extubatiuon
First NRS pain score (0-10 scale) at times of awakening | Intraoperative
  NRS (Numeric Rating Scale) Pain Score evaluated at times of awakening, evaluation from 0 (no pain) to 10 (worst imaginable pain) scale
First NRS pain score (0-10 scale) at arrival in PACU | Postoperative, evaluated at arrival in PACU
  First NRS Pain Score evaluated at arrival in PACU, evaluation from 0 (no pain) to 10 (worst imaginable pain)
NRS pain score (0-10 scale) at rest, in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  NRS Pain Score at rest, evaluated every 15 minutes until time for readiness for PACU discharge, evaluation from 0 (no pain) to 10 (worst imaginable pain)
NRS pain score (0-10 scale) with cough, in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  NRS Pain Score with cough, evaluated every 15 minutes until time for readiness for PACU discharge, evaluation from 0 (no pain) to 10 (worst imaginable pain)
NRS pain score (0-10 scale) on the Shoulder, in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  NRS Pain Score on the Shoulder, evaluated every 15 minutes until time for readiness for PACU discharge, evaluation from 0 (no pain) to 10 (worst imaginable pain)
Hydromorphone consumption (mg) in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  Total cumulative dose of titration of intravenous hydromorphone (mg), evaluated every 15 minutes until time for readiness for PACU discharge
PONV score (0-3 scale) in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  PONV (PostOperative Nausea and Vomiting) score, evaluated every 15 minutes until time for readiness for PACU discharge, evaluation from 0 (no nausea) to 3 (nausea and vomiting)
POSS score (1-4 scale) in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  POSS (Pasero Opioid-induced Sedation Scale) score evaluated every 15 minutes until time for readiness for PACU discharge, evaluation from 1 (awake and alert) to 5 (asleep deeply)
Respiratory depression number in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  Respiratory depression number evaluated every 15 minutes until time for readiness for PACU discharge
Blood pressure (mmHg) in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  Blood pressure (TAS/TAD/TAM) in mmHg evaluated every 15 minutes until time for readiness for PACU discharge
Time for PACU discharge based on Aldrete scores (0-10 scale), in PACU | Postoperative, evaluated every 15 minutes until time for PACU discharge
  Time for readiness for PACU discharge based on Aldrete scores (0-10), Aldrete score must be ≥ 9 for PACU discharge
NRS pain score (0-10 scale) at rest, evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  NRS Pain Score at rest, evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge, evaluation from 0 (no pain) to 10 (worst imaginable pain)
NRS pain score (0-10 scale) with cough, evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  NRS Pain Score with cough, evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge, evaluation from 0 (no pain) to 10 (worst imaginable pain)
NRS pain score (0-10 scale) on the Shoulder, evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  NRS Pain Score on the Shoulder, evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge, evaluation from 0 (no pain) to 10 (worst imaginable pain)
Hydromorphone consumption (mg), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Total cumulative dose of titration of intravenous hydromorphone (mg), evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge
Epidural consumption (mg), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Total cumulative dose of titration of epidural (mg), evaluated every day, from 24 hours postoperative until the cessation of the PCEA (Patient Controlled Epidural Analgesia)
PONV score (0-3 scale), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  PONV (PostOperative Nausea and Vomiting) score, evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge, evaluation from 0 (no nausea) to 3 (nausea and vomiting)
POSS score (1-4 scale), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  POSS (Pasero Opioid-induced Sedation Scale) score evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge, evaluation from 1 (awake and alert) to 5 (asleep deeply)
Respiratory depression number, evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Respiratory depression number evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge
Blood pressure (mmHg), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Blood pressure (TAS/TAD/TAM) in mmHg evaluated every day, from 24 hours postoperative until time for readiness for hospital discharge
Heart rate (bpm), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Heart rate (HR) in bpm (beats per minute), evaluated every day from 24 hours postoperative until time for readiness for hospital discharge
Oxygen saturation (%), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Oxygen saturation (SPO2) in %, evaluated every day from 24 hours postoperative until time for readiness for hospital discharge
Respiratory rate (bpm), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Respiratory rate (RR) in bpm (breaths per minute), evaluated every day from 24 hours postoperative until time for readiness for hospital discharge
Temperature (°C), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Temperature (T°C), evaluated every day from 24 hours postoperative until time for readiness for hospital discharge
Overall patient's satisfaction (0-100%), evaluated everyday from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Overall patient's satisfaction, evaluated every day from 24 hours postoperative until time for readiness for hospital discharge, evaluation from 0 (unsatisfied) to 100% (fully satisfied)
Quality of recovery (QoR-15), evaluated every day from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Patients' perceived quality of recovery (QoR-15). This questionnaire includes 15 questions that are divided into 2 parts, part A contains the first 10 questions that are scored between 0 (never) and 10 (constantly), and part B contains the last 5 questions scored between 0 (constantly) and 10 (never). Evaluation test every day from 24 hours postoperative until time for readiness for hospital discharge
6-minutes walking score, evaluated every day from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  6-minutes walking score. The object of this test is to walk as far as possible for 6 minutes in the hospital hallway. Six minutes is a long time to walk after this surgery type, so it's important to practise 6 Minute Walk every day on a flat hard surface. Evaluation test every day from 24 hours postoperative until time for readiness for hospital discharge
MOCA scores, evaluated every day from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  MOCA (Montreal Cognitive Assessment) scores test for Dementia, range from zero to 30, with a score of 26 and higher generally considered normal. In the initial study data establishing the MoCA, normal controls had an average score of 27.4, compared with 22.1 in people with mild cognitive impairment (MCI) and 16.2 in people with Alzheimer's disease.
  Evaluation test every day from 24 hours postoperative until time for readiness for hospital discharge
Time for first walking/mobilization, evaluated every day from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  The time for first walking/mobilization, consist to determine the precise moment when the patient is able to get up from his bed, and sit on a chair, with and without help
Time for first flatus, evaluated every day from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Determine the time of first flatus which are a sign of recovery of lower GI function
Time for return to food oral intake, evaluated every day from 24 hours postoperative to hospital | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Patient is able to tolerate at least one solid meal without nausea, vomiting, bloating or worsening abdominal pain. Patient drinks liquids actively (ideally > 800-1000 ml/day) and do not require intravenous fluids infusion to maintain hydration
Biological analysis, evaluated every day from 24 hours postoperative to hospital discharge | Evaluated 24 hours postoperative, then everyday until hospital discharge, an average of 21 days
  Biological analysis, intraoperative and daily during the 21 postoperative days: serum electrolytes (Na+ Cl- Ca2+ Ca total Phophore, glycemia) creatinine, DFG, CRP, hemoglobin, white blood cell and platelet counts, serum albumin, INR, PTT
Rate of hospital readmission and mortality postoperative | Postoperative evaluation, up to 30 days following surgery
  Rate of hospital readmission and mortality postoperative up to 30 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PR Richebé, MD PhD, Principal Investigator — CIUSSS Est de l'île de Montréal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal East, Quebec, Canada